CLINICAL TRIAL: NCT05007288
Title: A Single Center Evaluation of Restorative Eye Treatment and Inhance With Trihex Technology Effects on the Aesthetic Outcomes When Used Pre and Post Upper Blepharoplasty
Brief Title: Restorative Eye Treatment and INhance in Upper Eyelid Blepharoplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Professor of Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200939
Record Dates: First submitted 2021-05-11; First posted 2021-08-16 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Eyelid Dermatochalasis; Dermatochalasis
Keywords: Blepharoplasty
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RET Treated Eye Plus INhance Group (Experimental): Participants randomized to receive the restorative eye treatment (RET) intervention on either the left or right eyelid will administer the RET cream on the eyelid daily for 4 consecutive weeks prior to scheduled standard of care (SOC) blepharoplasty. After surgery, participants will receive INhance with Trihex technology applied to both eyelids daily for 10 consecutive days post surgery.
  Interventions: Other: Restorative Eye Treatment (RET) cream; Other: INhance with Trihex Technology
- RET Untreated eye Plus INhance Group (Experimental): Participants randomized to not receive the RET intervention will not receive any intervention prior to scheduled standard of care (SOC) blepharoplasty. After surgery, participants will receive INhance with Trihex technology applied to both eyelids daily for 10 consecutive days post surgery.
  Interventions: Other: INhance with Trihex Technology

INTERVENTIONS:
Other: Restorative Eye Treatment (RET) cream — RET cream will be applied topically to either the left of right eyelid once daily for 4 consecutive weeks.
  Arms: RET Treated Eye Plus INhance Group
Other: INhance with Trihex Technology — INhance will be applied topically to both eyelids once daily for 10 consecutive days after the SOC blepharoplasty surgery.

SUMMARY:
The purpose of this research is to determine if restorative eye treatment (RET) and Inhance with trihex technology used before and after blepharoplasty can lead to better skin quality before undergoing blepharoplasty, and if these products will lead to less visible scarring and faster healing after blepharoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who are about to have blepharoplasty at the Bascom Palmer Eye Institute by Dr. Wendy Lee.
2. Men and women with no known medical conditions that, in the investigator's opinion, may affect wound healing and interfere with study participation (e.g. diabetes, skin disorder etc.).
3. Participants willing to provide consent for photographic release.
4. Participants must not be using any new skincare products, other than the study products provided, on the treatment area for the duration of the study.
5. Participants willing to avoid extended periods of sun exposure and all use of tanning beds for the duration of the study.
6. Participants must be willing to refrain from any other treatments or procedures to the treatment area during the duration of the study.
7. 18 years old or older.

Exclusion Criteria:

1. Any dermatological disorder or poor health, which in the investigator's opinion, may interfere with the accurate evaluation of the participants' skin characteristics or inhibit wound healing.
2. Participants who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
3. Participants that have been using topical products around their upper or lower eyes within 30 days.
4. Participants who are, in the opinion of the investigator, unwilling or unable to comply with the requirements of the protocol.
5. Pregnant or lactating participants will be excluded, as well as participants planning on becoming pregnant during the study duration.
6. Participants with recent excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing).
7. A participant with a history of keloids or hypertrophic scars.
8. Participants known to harbour a blood borne disease (e.g. Hepatitis A Virus (HAV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV ), HIV)
9. Special populations: Prisoners, Pregnant women, Adults unable to consent, Individuals who are not yet adults.
10. Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Collagen Content | Up to 1 month prior to blepharoplasty surgery
  Assessed from eyelid tissue samples
Elastin Content | Up to 1 month prior to blepharoplasty surgery
  Assessed from eyelid tissue samples
Post operative bruising | Up to 2 weeks post blepharoplasty surgery
  Bruising will be assessed on a 1-5 scale with the higher score indicating more bruising.

SECONDARY OUTCOMES:
Post operative swelling | Up to 2 weeks post blepharoplasty surgery
  Swelling will be assessed on a 1 to 5 scale with the higher score indicating more swelling

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W Lee, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reivitis A, Karimi K, Griffiths C, Banayan A. A single-center, pilot study evaluating a novel TriHex peptide- and botanical-containing eye treatment compared to baseline. J Cosmet Dermatol. 2018 Jun;17(3):467-470. doi: 10.1111/jocd.12542. Epub 2018 Apr 16. PMID 29663676
- [Result] Widgerow AD, Jacob C, Palm MD, Garruto JA, Bell M. Developing a Topical Adjunct to Injectable Procedures. J Drugs Dermatol. 2020 Apr 1;19(4):398-404. doi: 10.36849/JDD.2020.5016. PMID 32272517
- [Result] Widgerow AD, Jiang LI, Calame A. A single-center clinical trial to evaluate the efficacy of a tripeptide/hexapeptide antiaging regimen. J Cosmet Dermatol. 2019 Feb;18(1):176-182. doi: 10.1111/jocd.12507. Epub 2018 Mar 4. PMID 29504212